CLINICAL TRIAL: NCT04617145
Title: Impact of Aerobic Versus Resistive Training on Functional Capacity in Acute Myeloid Leukemia Survivors; a Comparative Study
Brief Title: Aerobic Versus Resistive Training on Functional Capacity in Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA201918
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia in Remission
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: parallel randomized single blinded study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Active Comparator): Included 30 patients who underwent aerobic training with 50 %-60% of maximum heart rate in the form of cycling by Bicycle ergometer for eight weeks, three sessions/week.
  Interventions: Other: Aerobic exercise
- Resistive exercise group (Active Comparator): Included 30 patients who underwent a resistive training which were conducted in the form of a series of exercises using free weights, and dumbles to increase the strength of arms, pectoral muscles, abdominal, back muscles and gluteal region. Sessions were conducted three sessions/week for eight weeks.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — resistive training which were conducted in the form of a series of exercises using free weights, and dumbles to increase the strength of arms, pectoral muscles, abdominal, back muscles and gluteal region. Patients carried out three sets of 20-30 dynamic repetitions or static isometric exercises for 40-60 seconds for each muscle group and rested 1-2 min between series. Sessions were conducted three sessions/week for eight weeks.
  Other Names: Resistive exercise

SUMMARY:
Sixty patients with AML from both sexes aged from 35-45 years were selected from hematology department in Nasser Institute Hospital where the study was conducted. Patients were randomly assigned into two groups equal in number. Group (A) underwent aerobic exercises in the form of cycling with 50-60% of maximum heart rate. Group (B) underwent resistive training conducted in the form of a series of exercises using free weights, and dumbles. Sessions were conducted three times /week for eight weeks. Six minutes' walk test (6MWT), 10 repetitions maximum test (10 RM), ventilatory function test, fatigue and quality of life (QOL) scales were used to assess functional capacity in both groups.

DETAILED DESCRIPTION:
Aerobic Ex Group: Included 30 patients who underwent aerobic training with 50 %-60% of maximum heart rate in the form of cycling by Bicycle ergometer for eight weeks, three sessions/week.

Resistive Ex Group: Included 30 patients who underwent a resistive training which were conducted in the form of a series of exercises using free weights, and dumbles to increase the strength of arms, pectoral muscles, abdominal, back muscles and gluteal region. Patients carried out three sets of 20-30 dynamic repetitions or static isometric exercises for 40-60 seconds for each muscle group and rested 1-2 min between series. Sessions were conducted three sessions/week for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia survivors from both sexes
* Their age ranged from 35-45 years.
* Patients were in remission stage contains less than 5% blast cells in their bone marrow, absolute neutrophil count (>1000/microL), platelet count(>100,000/microL),and independence from red cell transfusion.

Exclusion Criteria:

* Extramedullary leukemia
* musculoskeletal deformities
* severe anemia (hemoglobin less than 8g/dl).
* Autoimmune thrombocytopenia (platelets less than 10000UL or leucocytes count more than 3000UL).

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Six minutes walking Distance | It is performed before and after the study(8 weeks interval) for both groups
  which used to measure the distance the patient was able to walk over a total of six minutes According to American thorax society guidelines; patients were instructed to walk as fast as long as possible , in a 30 meters obstacle free corridor limited by turnaround cones and distance was calculated
10 repetition maximum test | It is performed before and after the study(8 weeks interval) for both groups
  which the greatest amount of weight a person can lift number of times. The amount of weight that can be lifted exactly 10 times is 10 RM
Vital capacity | It is performed before and after the study(8 weeks interval) for both groups
  was measured by using electronic spirometry used to conduct ventilatory function testing

SECONDARY OUTCOMES:
Maximum oxygen consumption | It is performed before and after the study(8 weeks interval) for both groups
  Results of (6MWT) was used to calculate Vo2 max by using Cahalin equation as follows; Vo2 max = 0.03x distance in meters +3.98, in which distance is obtained from (6MWT)
Fatigue assessment scale (FAS) | It is performed before and after the study(8 weeks interval) for both groups
  FAS is a 10-item scale evaluating symptoms of chronic fatigue
Quality of life questionnaire (QOL) | It is performed before and after the study(8 weeks interval) for both groups
  was used to evaluate the quality of life before and after training for both groups.The Quality of Life Instrument (CANCER PATIENT/CANCER SURVIVOR VERSION) is a forty one-item ordinal scale. The scoring should be based on a scale of 0 = worst outcome to 10 = best outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No